CLINICAL TRIAL: NCT00004157
Title: Combination of Interleukin 11 (Neumega) With G-CSF to Mobilize Autologous Peripheral Blood Stem Cells (PBSC)
Brief Title: Interleukin-11 Plus Filgrastim Prior to Peripheral Stem Cell Transplantation in Patients With Non-Hodgkin's Lymphoma, Hodgkin's Disease, Breast Cancer, or Other Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1365.00; FHCRC-1365.00; NCI-G99-1622; CDR0000067395 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-12-10; First posted 2004-02-12 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer; Gestational Trophoblastic Tumor; Kidney Cancer; Lymphoma; Neuroblastoma; Ovarian Cancer; Sarcoma; Testicular Germ Cell Tumor
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; recurrent adult Hodgkin lymphoma; recurrent childhood rhabdomyosarcoma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; recurrent childhood lymphoblastic lymphoma; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent ovarian germ cell tumor; ovarian yolk sac tumor; ovarian embryonal carcinoma; ovarian polyembryoma; ovarian choriocarcinoma; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian mixed germ cell tumor; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; poor prognosis metastatic gestational trophoblastic tumor; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; previously treated childhood rhabdomyosarcoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Breast Neoplasms; Gestational Trophoblastic Disease; Kidney Neoplasms; Lymphoma; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Testicular Germ Cell Tumor; Hodgkin Disease; Carcinoma, Ovarian Epithelial; Wilms Tumor; Testicular Neoplasms; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Seminoma; Carcinoma, Embryonal; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Interleukin-11

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interleukin-11

SUMMARY:
RATIONALE: Interleukin-11 and filgrastim stimulate the production of blood cells. Giving these drugs to stimulate peripheral stem cells that can be collected for peripheral stem cell transplantation may result in fewer side effects after transplant.

PURPOSE: Phase II trial to study the effectiveness of interleukin-11 plus filgrastim prior to peripheral stem cell transplantation in patients who have non-Hodgkin's lymphoma, Hodgkin's disease, breast cancer, or other solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the tolerability of interleukin-11 (IL-11) with filgrastim (G-CSF) in patients with non-Hodgkin's lymphoma, Hodgkin's disease, breast cancer, or other solid tumors. II. Evaluate the ability to collect CD34 cells and the number of apheresis collections required to reach the target number of CD34 cells in this patient population. III. Evaluate the time to recovery of platelets and neutrophils and the number of platelet and red blood cell transfusions required following IL-11 and G-CSF mobilized peripheral blood stem cell infusion in these patients.

OUTLINE: Patients receive interleukin-11 (IL-11) subcutaneously (SQ) on days 1-10 and filgrastim (G-CSF) SQ on days 4-10. Patients undergo peripheral blood stem cell (PBSC) collection on days 7-10 until the target number of cells is achieved or for a maximum of 4 collections. Patients are followed until transplantation.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of non-Hodgkin's lymphoma, Hodgkin's disease, breast cancer, or other solid tumors with eligibility for FHCRC/PSOC protocols involving autologous peripheral blood stem cell transplantation No evidence of bone marrow disease No pericardial effusion, pleural effusion, or ascites No CNS involvement Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 70 and under Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.5 times upper limit of normal (ULN) SGOT no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL No medically unmanageable, severe hypokalemia Cardiovascular: No history of atrial arrhythmia or congestive heart failure No history of thromboembolic disease, except successfully treated catheter related thrombosis LVEF at least 45% Other: No active infection requiring systemic antibiotics HIV negative No known allergy to murine or E. coli proteins No documented prior anaphylactic reaction to interleukin-11 or filgrastim (G-CSF) No papilledema No history of Factor V Leiden defect, factor II, antithrombin III, Protein C or Protein S deficiencies Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: No prior cumulative dose of doxorubicin greater than 300 mg/m2 At least 3 weeks since prior chemotherapy Endocrine therapy: No concurrent estrogen supplementation Radiotherapy: No prior radiotherapy to the pelvic area Surgery: Not specified Other: No chronic diuretic therapy At least 1 week since prior aspirin or anticoagulants except low dose anticoagulation to prevent catheter thrombosis

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States